CLINICAL TRIAL: NCT06793683
Title: Early Detrusor Chemodenervation to Preserve Bladder Compliance and Longevity After Spinal Cord Injury
Brief Title: Early BOTOX After Spinal Cord Injury
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Claire Yang, MD, Professor: Department of Urology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00018758
Record Dates: First submitted 2024-12-06; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries
Keywords: SCI; Neurogenic Bladder; Chemodenervation with BoNT-A; Botox; Autonomic Dysreflexia
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic; Autonomic Dysreflexia | interventions — Botulinum Toxins, Type A; Sodium Chloride; Injections

STUDY DESIGN:
Intervention Model Description: The investigators hope to recruit 10 participants randomly assigned to 7 cases (those that will receive Botox bladder injections) and 3 controls (those that will receive placebo bladder injections).
Who Masked: Participant
Masking Description: Participants will be blinded during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bladder Chemodenervation (Botox) Injection Procedure (Active Comparator): BoNT-A (Botox) 200 U, will be injected into the detrusor (bladder wall muscle).
  Interventions: Drug: Bladder chemodenervation (Botox)
- Bladder Sham (saline) Injection Procedure (Sham Comparator): Saline will be injected into the detrusor (bladder wall muscle).
  Interventions: Procedure: Bladder Sham (Saline) Injection Procedure

INTERVENTIONS:
Drug: Bladder chemodenervation (Botox) — BoNT-A (Botox) 200 U will be injected into the detrusor (bladder wall muscle).
  Arms: Bladder Chemodenervation (Botox) Injection Procedure
Procedure: Bladder Sham (Saline) Injection Procedure — 20mL placebo (saline only), will be injected into the detrusor (bladder wall muscle).
  Arms: Bladder Sham (saline) Injection Procedure

SUMMARY:
The investigators would like to improve our understanding of how early intervention with the use of bladder chemodenervation can preserve bladder function in those with a new SCI. Although detrimental cystometric and tissue changes are known to occur, often within 3 months after SCI, the investigators seek to document the time course of these changes and the range of severity of those changes in both those participants that receive prophylactic treatment and those who do not.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-65 years of age at time of SCI.
* English speaking
* Recent SCI (within 20 weeks of injury).
* Documentation of a spinal cord injury at T6 or higher, American Spinal Injury Association Impairment Scale (AIS) level A or B as designated on initial (72 hour) AIS exam.
* Ability for subject to comply with the requirements of the study.
* Written informed consent obtained from subject.

Exclusion Criteria:

* Inability to return to research site (Harborview Medical Center) for follow-up studies after initial hospitalization.
* Acute (as part of concurrent hospitalization) or history of bladder surgery (urethral or prostate surgery acceptable) or injury.
* Inability to provide informed consent.
* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Incarcerated in a detention facility or in police custody.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Active medical problems precluding the safe conduct of urodynamics, bladder chemodenervation, bladder biopsy (e.g., evidence of active bladder infection, ruled out by urine culture prior to procedures)
* Known hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation
* Cardiovascular instability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-27 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Enrollment goals | Each participant will be evaluated for a period of up to 12 months after the time of enrollment.
  Outcomes of this pilot trial will provide human data on the feasibility of recruiting 10 participants into a randomized study of early chemodenervation.
  The enrollment goal is 10 participants who will complete the 12-month study protocol.
  If ≥ 8 participants complete the protocol, it will be considered feasible. If ≤ 5 participants complete the protocol, it will be considered unfeasible. If 6-7 participants complete the study, it will be considered indeterminate.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | For each participant any AE's will be documented, at time of AE, beginning at study enrollment and throughout each participants 12 month enrollment period.
  Patients will be monitored for adverse events as a result of the procedures.
  * Evidence of Urinary Tract Infections
  * Hematuria
  * Anesthesia Complications
  Any adverse events (AE) will be graded 1 through 5, with unique clinical descriptions of severity for each AE, based upon the AE guidelines as published in the CAE v4.0

SECONDARY OUTCOMES:
Variance of measurements for functional data | Variances of all measurements and data, for each subject, will be analyzed at the conclusion of their study participation, 12 months post enrollment.
  Determination of variance of measurements for functional data, including:
  Cystometric values will be analyzed as a continuous variable and compared between early detrusor oBoNT-A injected cases and controls at the 6- and 12-month time points. Standard clinical care characterizes bladder compliance as poor for values <10 mL/cm H2O, indeterminate for values between 10 mL/cm H2O and 20 mL/cm H2O, and good for values >20 mL/cm H2O. To interpret our data, we will use these existing clinical guidelines in concert with statistical differences that arise.
Variance of measurements for histological data | Variances of all measurements and data will be analyzed at the conclusion of the study (expected in 2028).
  Determination of variance of measurements for histological data, including:
  Histological analyses of the bladder biopsy samples will include standard histological staining to evaluate hypertrophy and fibrosis, and how these parameters change with time (baseline, 6 months and 12 months post SCI).

CONTACTS AND LOCATIONS:
Overall Officials: Claire C Yang, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Comperat E, Reitz A, Delcourt A, Capron F, Denys P, Chartier-Kastler E. Histologic features in the urinary bladder wall affected from neurogenic overactivity--a comparison of inflammation, oedema and fibrosis with and without injection of botulinum toxin type A. Eur Urol. 2006 Nov;50(5):1058-64. doi: 10.1016/j.eururo.2006.01.025. Epub 2006 Feb 6. PMID 16517054
- [Background] Ginsberg D, Gousse A, Keppenne V, Sievert KD, Thompson C, Lam W, Brin MF, Jenkins B, Haag-Molkenteller C. Phase 3 efficacy and tolerability study of onabotulinumtoxinA for urinary incontinence from neurogenic detrusor overactivity. J Urol. 2012 Jun;187(6):2131-9. doi: 10.1016/j.juro.2012.01.125. Epub 2012 Apr 12. PMID 22503020
- [Background] Ku JH, Choi WJ, Lee KY, Jung TY, Lee JK, Park WH, Shim HB. Complications of the upper urinary tract in patients with spinal cord injury: a long-term follow-up study. Urol Res. 2005 Dec;33(6):435-9. doi: 10.1007/s00240-005-0504-4. Epub 2005 Nov 30. PMID 16317536
- [Background] Janzen J, Vuong PN, Bersch U, Michel D, Zaech GA. Bladder tissue biopsies in spinal cord injured patients: histopathologic aspects of 61 cases. Neurourol Urodyn. 1998;17(5):525-30. doi: 10.1002/(sici)1520-6777(1998)17:53.0.co;2-f. PMID 9776015
- [Background] Bywater M, Tornic J, Mehnert U, Kessler TM. Detrusor Acontractility after Acute Spinal Cord Injury-Myth or Reality? J Urol. 2018 Jun;199(6):1565-1570. doi: 10.1016/j.juro.2018.01.046. Epub 2018 Jan 17. PMID 29352989
- [Background] Rosier PFWM, Valdevenito JP, Smith P, Sinha S, Speich J, Gammie A; Members of the ICS Working Group PFS23. ICS-SUFU standard: Theory, terms, and recommendations for pressure-flow studies performance, analysis, and reporting. Part 1: Background theory and practice. Neurourol Urodyn. 2023 Nov;42(8):1590-1602. doi: 10.1002/nau.25192. Epub 2023 Apr 25. PMID 37096828
- [Background] Welk B, Morrow S, Madarasz W, Baverstock R, Macnab J, Sequeira K. The validity and reliability of the neurogenic bladder symptom score. J Urol. 2014 Aug;192(2):452-7. doi: 10.1016/j.juro.2014.01.027. Epub 2014 Feb 8. PMID 24518764
- [Background] Tang DH, Colayco D, Piercy J, Patel V, Globe D, Chancellor MB. Impact of urinary incontinence on health-related quality of life, daily activities, and healthcare resource utilization in patients with neurogenic detrusor overactivity. BMC Neurol. 2014 Apr 4;14:74. doi: 10.1186/1471-2377-14-74. PMID 24708598
- [Background] Bushnell JY, Cates LN, Hyde JE, Hofstetter CP, Yang CC, Khaing ZZ. Early Detrusor Application of Botulinum Toxin A Results in Reduced Bladder Hypertrophy and Fibrosis after Spinal Cord Injury in a Rodent Model. Toxins (Basel). 2022 Nov 10;14(11):777. doi: 10.3390/toxins14110777. PMID 36356027